CLINICAL TRIAL: NCT06286930
Title: Cerebellar tDCS Stimulation in Children and Adult Women With Anorexia Nervosa Disorder- A Pilot Study
Brief Title: Cerebellar tDCS Stimulation in Children and Adult Women With Anorexia Nervosa Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Carrie McAdams, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2023-0470
Record Dates: First submitted 2024-01-29; First posted 2024-02-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Anorexia Nervosa
Keywords: transcranial direct current stimulation; Adolescents; Adults; tDCS
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- anodal tDCS, then cathodal tDCS (Experimental): Participants receive 1, 20-minute anodal tDCS stimulation. After a washout period of 2-3 weeks, then receive 1, 20-minute cathodal tDCS stimulation.
  Interventions: Device: anodal trans cranial direct current stimulation (tDCS); Device: cathodal trans cranial direct current stimulation (tDCS)
- cathodal tDCS, then andoal tDCS (Experimental): Participants receive 1, 20-minute cathodal tDCS stimulation. After a washout period of 2-3 weeks, then receive 1, 20-minute anodal tDCS stimulation.
  Interventions: Device: anodal trans cranial direct current stimulation (tDCS); Device: cathodal trans cranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: anodal trans cranial direct current stimulation (tDCS) — 1 20-minute anodal tDCS stimulation
Device: cathodal trans cranial direct current stimulation (tDCS) — 1 20-minute cathodal tDCS stimulation

SUMMARY:
Hypothesis: Will the use of tDCS brain modulation in the cerebellum assist in restricted behaviors, social cognition and cognitive flexibility in women with anorexia nervosa in addition to other therapies?

Primary Outcomes:

1. To observe the impacts and outcomes of cerebellar transcranial direct current stimulation (tDCS) on social behaviors measured by Cyberball and Trust Game.
2. To observe the neuropsychological impacts of cerebellar tDCS through fMRI imaging as well as looking at the Region of Interest (ROI) of changes in the Default Mode Network and Cerebellum circuits and their activation levels in those networks.

Secondary Outcomes:

1.To observe the impacts and outcome of cerebellar transcranial direct current stimulation (tDCS) measuring the differences between anodal and cathodal stimulation. To observe potential increases in responses to social stimuli, decreases in eating disorder/depressive symptomology via cathodal stimulation. To also observe potential little to no changes in social stimuli and eating disorder/depressive symptomology via anodal stimulation.

DETAILED DESCRIPTION:
The study will be randomized, single blind design. It will involve a group of 15 female participants ranging in the ages of 15-30 years old diagnosed with Anorexia Nervosa. Diagnosis will be confirmed by recruitment methods of in-clinic referrals. Each participant will undergo the two different electrode stimulations of the tDCS. Each participant will get anodal and cathodal stimulation. The participants will be unaware of which one they are getting during stimulation, but the researcher will be informed of which stimulation is occurring. The participant will receive 1mA stimulation of the tDCS for 20 minutes in the MRI scanner. After the stimulation is complete in the scanner, the participant will be asked to complete tasks in the scanner as well. The study involves initial screening to determine eligibility to participate. Once eligibility criteria is met, the participant will sign consent via DocUSign. After this virtual visit is complete, the participant will be asked to come in for intake visit. At the intake, the participant will undergo a series of questionnaires and tasks to complete as part of pre-scanning. The next session will be stimulation and MRI imaging. Participant will undergo resting state and a structural scan. After the scans are complete, the participant will receive 20 minutes of tDCS stimulation. After the simulation is complete the participant will be asked to engage in tasks in the scanner. Finally, after the scanning session, the participant will come back for a post session that is the same as the intake and undergo questionnaires and tasks to complete. After the post session, researchers will reach out to participants one week and one month after MRI imaging to go over safety questionnaire of the tDCS. The participant will have a total of 5 sessions which may include both in-person and/or virtual visits with screening session, first session, second session, one week follow-up session, and one-month follow-up session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Anorexia Nervosa (AN)
* Female participants
* Age 15-30 years old inclusive at time of enrollment
* Ability of parent or legal guardian to provide informed consent if participant is under 18 years old.
* Ability of patients ages 15-17 to give assent to the study.
* Completion of the signed HIPAA authorization form by a parent or legal guardian or by participants (18 years of age).

Exclusion Criteria:

* Pregnancy
* Known history of traumatic brain injury that required medical care
* Non-English speaking (based on standardized neuropsychological testing and questionnaires)
* Claustrophobic
* Brain Implants
* Pacemakers
* Hearing or visual impairment
* Any biomedical or metal implants in any part of the body (excluding orthopedic implants)

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Must be female/ biologically female
Enrollment: 15 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
tDCS impact on social behaviors using Cyberball | 1 year
  To observe the impacts and outcomes of cerebellar transcranial direct current stimulation (tDCS) on social behaviors measured by Cyberball. Cyberball is a virtual ball toss game utilized to measure ostracism, social exclusion, rejection, etc. This measure predicts whether or not the behavior of the participant will change how they react to the game after receiving transcranial direct current stimulation (tDCS).
tDCS impact on social behaviors using the Trust Game | 1 year
  To observe the impacts and outcomes of cerebellar transcranial direct current stimulation (tDCS) on social behaviors measured by the Trust Game. The Trust Game Examines how expectations about prior behaviors influence current behavior and responses. Using a computational psychiatry approach in which neuroimaging data is sorted based on the behaviors experienced in the game (reciprocity). The prediction is to see after tDCS administration, will the behaviors of the participant change towards the online player in the trust game or not.
neurological impacts of tDCS as measured by fMRI imaging | 1 year
  To observe the potential re-connection between the cerebellum and the default mode network as well as other areas of the brain during transcranial direct current stimulation measured by fMRI imaging.

SECONDARY OUTCOMES:
measure the differences of social stimuli and eating disorder/depressive symptomology | 1 year
  To observe potential increases in responses to social stimuli, decreases in eating
  disorder/depressive symptomology via transcranial direct current stimulation.
measure the differences of social stimuli and eating disorder/depressive symptomology | 1 year
  To observe potentially little to no changes in social stimuli and eating disorder/depressive symptomology via transcranial direct current stimulation.
measuring the differences of social stimuli and eating disorder/depressive symptomology measuring using the Food Rating Task. | 1 year
  After receiving transcranial direct current stimulation, it is predicted that after stimulation, there will be differences in how the participant will choose certain food items. It suggests that the experience of tastiness changes over time and may contribute to perpetuation of anorexia nervosa.
measure the differences of social stimuli and mental flexibility with Trail Making Task | 1 year
  To observe after transcranial direct current stimulation, if there are differences in mental flexibility with participants with anorexia nervosa. The Trail Making Task A is a measure of simple visual attention, scanning, and psychomotor speed. In contrast, Trail Making Task B is a measure of complex/divided visual attention, and mental flexibility.
measure the differences of social stimuli and eating disorder/depressive symptomology utilizing Patient Health Questionnaire-9. | 1 year
  To observe the differences in self-report answers after stimulation.PHQ-9 observes depression severity.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Multispecialty Psychiatry Clinic, Dallas, Texas, United States